CLINICAL TRIAL: NCT05451030
Title: The Effect of Remote Ischemic Preconditioning on Cerebral Circulation Time in Patients With Severe Carotid Artery Stenosis (RIP-CCT): A Prospective, Randomized Controlled, Blind Outcome Evaluation, Multi-center Study
Brief Title: Effect of Remote Ischemic Preconditioning on Cerebral Circulation Time in Patients With Severe Carotid Artery Stenosis (RIP-CCT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Hui-Sheng Chen, Head of Neurology, General Hospital of Shenyang Military Region
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Y (2022) 022
Record Dates: First submitted 2022-07-05; First posted 2022-07-11 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Carotid Artery Stenosis
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- remote ischemic preconditioning (Experimental)
  Interventions: Device: remote ischemic preconditioning
- control group (Sham Comparator)
  Interventions: Device: remote ischemic preconditioning

INTERVENTIONS:
Device: remote ischemic preconditioning — The cuff of a pneumatic electronic auto-control device placed around the bilateral upper limbs was used to deliver the protocol: 5 cycles of cuff inflation (200mmHg for 5 minutes) and deflation (for 5 minutes), for a total procedure time of 50 minutes, twice daily from the first DSA to the day of carotid artery stenting.

SUMMARY:
Cerebral circulation time in patients with severe carotid artery stenosis was found to be associated with hyperperfusion syndrome. Remote ischemic preconditioning can change the ability of cerebral autoregulation. The prospective, randomized controlled, blind outcome evaluation, multi-center study aimed to investigate the effect of remote ischemic preconditioning on cerebral circulation time in patients with severe carotid artery stenosis.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older, regardless of gender;
* patients with severe carotid stenosis eligible for stenting (70-99% stenosis confirmed by DSA);
* non-responsible vessel stenosis <50% if bilateral carotid stenosis or combined posterior circulation stenosis is present;
* first DSA suggestive of ≥ 0.8 seconds difference (CCT on the affected side - CCT on the healthy side);
* baseline modified Rankin Scale (mRS) ≤ 2 points.
* signed the informed consent form.

Exclusion Criteria:

* baseline mRS ≥ 3 points;
* severe long-segment calcification of the carotid artery, severe distortion of aortic arch branches, anatomical variation of the aortic arch, and etc, which are not suitable for stenting
* spontaneous intracranial hemorrhage within 12 months;
* previous severe stroke or myocardial infarction within 3 months;
* active bleeding and coagulation disorders, which is contraindication to heparin and antiplatelet agents;
* a large intracranial aneurysm that cannot be treated simultaneously;
* severe insufficiency of vital organs such as the heart, lungs, liver and kidneys, or malignant tumors with an expected survival cycle of less than six months;
* total occlusion of carotid artery without obvious cerebral ischemic symptoms
* unable to tolerate anesthesia;
* severe dementia;
* uncontrolled hypertension ;
* allergy to contrast media;
* pregnancy;
* being involved in studies with other drugs or instruments, etc;
* contraindications to remote ischemic preconditioning, such as those with more severe soft tissue injuries, fractures or vascular injuries in the upper extremity, or peripheral vascular lesions in the distal upper extremity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2022-06-28 (Actual); Primary Completion 2023-03-06 (Actual); Study Completion 2023-03-06 (Actual)

PRIMARY OUTCOMES:
Changes in cerebral circulation time | pre-intervention

SECONDARY OUTCOMES:
changes in contrast staining on brain computerized tomography after carotid artery stenting | 1 hours and 24 hours after carotid artery stenting
changes in collateral scoring based on digital subtraction angiography | pre-intervention
occurence of hyperperfusion syndrome after carotid artery stenting | 24 hours and 7 days after carotid artery stenting

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, General Hospital of Northern Theater Command, Shenyang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Liu QY, Cui Y, Li W, Qiu J, Nguyen TN, Chen HS. Effect of remote ischemic preconditioning on cerebral circulation time in severe carotid artery stenosis: Results from the RIC-CCT trial. Cell Rep Med. 2024 Nov 19;5(11):101796. doi: 10.1016/j.xcrm.2024.101796. Epub 2024 Oct 28. PMID 39471820